CLINICAL TRIAL: NCT07380698
Title: The Effect of Dose and Storage Conditions of Indocyanine Green on Efficacy and Cost in Sentinel Lymph Node Mapping in Gynecological Cancer
Acronym: DOSTCONICG
Status: Recruiting | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ghanim Khatib, Associated Professor, Cukurova University
Other Study IDs: 159/24
Record Dates: First submitted 2026-01-01; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer; Vulvar Cancers; Cervical Cancer; Indocyanine Green (ICG)
Keywords: endometrial cancer; vulvar cancers; cervical cancers
MeSH Terms: conditions — Endometrial Neoplasms; Vulvar Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research will determine the impact of optimizing dosage and storage conditions for indocyanine green on health outcomes and will contribute to improving treatment processes in gynecological cancers. Ultrastaging will increase the detection of micrometastases. Furthermore, the cost impact of these optimizations will be evaluated. It will help develop more effective, safe, and cost-effective methods for sentinel lymph node mapping in gynecological cancers. Furthermore, significant savings in healthcare costs could be achieved.

DETAILED DESCRIPTION:
Indocyanine Green (ICG) is a substance used in many areas of medicine, particularly in surgical procedures for vascular imaging, organ function assessment, and the treatment of various types of cancer. In recent years, this substance has also gained significant ground in gynecological cancers. The use of indocyanine green in gynecological cancers is particularly notable for its role in identifying cancer cells, performing lymph node biopsies, and performing minimally invasive surgeries.

Indocyanine green has become an important tool in the treatment of gynecological cancers, particularly in lymph node biopsies and minimally invasive surgeries. Its applications are increasingly expanding as it helps identify the path of cancer spread and enhances surgical precision. This substance allows surgeons to perform more accurate and effective interventions while also accelerating patient recovery.

Sentinel lymph node (SLN) mapping is increasingly used in gynecologic cancers as a less morbid staging method, an alternative to systematic pelvic and para-aortic lymphadenectomy. Numerous prospective studies have demonstrated the accuracy and reliability of the SLN technique, particularly in endometrial, cervical, and vulvar cancers. Indocyanine green (ICG), when used in conjunction with near-infrared fluorescence imaging, has become the most frequently used method due to its high sensitivity and bilateral detection rate.Patients diagnosed with endometrial, cervical, and vulvar cancer and scheduled for SLN mapping will be included in the study; potential confounding variables such as patient characteristics (age, BMI, comorbidities), tumor characteristics (histology, stage), surgical approach, and surgeon experience will also be considered in the analyses. Indocyanine green administration in gynecological cancers:

1. Standard dose (1.25 mg/mL, 4 x 1 mL)
2. A low-volume protocol (1 mL) may be tried in low-risk cases for minimal intervention, but signal may be reduced.
3. A high-volume application (8-10 mL) may be preferred in obese or signal-deficient patients; signal strength may be increased.
4. A high concentration (2.5 mg/mL) has been found effective in some studies, but should be used with caution due to the risk of suppressing ICG's own fluorescence.

Standard storage conditions:

Storage at 2-8°C (refrigerated) in dark glass vials protected from light and moisture.

Short-term storage at room temperature (15-25°C) after preparation is suitable. Use within 24 hours is recommended. In this study, sentinel lymph node mapping will be performed by injecting 1 cc of indocyanine green diluted with sterile water (25 mg + 20 mL water → 1.25 mg/mL) into the submucosa of the cervical os at the 3-9 o'clock positions.

Prepared ICGs will be stored in a dark environment at +4°C.

The data obtained will evaluate the effects of the dosage on mapping success and also reveal the potential effects of indocyanine green storage conditions on efficacy and cost. This study aims to contribute to the development of a safer, more effective, and more economical mapping method for gynecological cancers.

Parameters used in this study:

* Age (years)
* BMI (kg/m²)
* Parity
* Comorbidities (DM, HT, cardiac/AKI, COPD, renal failure)
* Drug/allergy history (especially iodine/ICG/green dye)
* Previous pelvic surgery/lymph node dissection/RT-CT history
* ASA score
* Cancer type: endometrium, cervix, vulva
* Cancer stage (clinical and/or pathological)
* Histology (endometrioid/serous/clearcell/squamous, etc.)
* Tumor size (mm), depth of myometrial invasion (%) in endometrial cancers, LVSI (present/absent), depth of stromal invasion in cervical tumors, parametrial involvement, lesion location and size in the vulva
* Need for reinjection: Present/Absent
* Injection sites and plan: 3-9 line (superficial/deep) on the cervix, clitoris level on the vulva, labia majora; cervical injection standardization for the endometrium. -Storage conditions
* Freshly prepared vs. stored for a certain period
* Temperature: Room temperature vs. Refrigerator
* Operative: Laparoscopic/Laparotomic
* Operative duration (min), time to SLN (min)
* Intraoperative complications (allergic reaction, tissue staining problems, etc.)
* Number of lymph nodes: Total SLNs removed, SLNs per side
* Anatomical distribution: Obturator, external/internal iliac, parametrial, presacral, etc.
* Micro/macrometastasis, isolated tumor cells

ELIGIBILITY:
Inclusion Criteria:

* cervical cancer, endometrial cancer, vulvar cancer, using indocyanine green, sentinel lymph node dissection

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Women who have endometrial or cervical or vulvar cancer
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2026-08-03 (Estimated); Study Completion 2026-09-03 (Estimated)

PRIMARY OUTCOMES:
Sentinel lymph node detection success rate associated with optimized indocyanine green (ICG) dosage and storage conditions. | Baseline (pre-procedure), perioperative/periprocedural period, and up to 24 weeks post-procedure.

SECONDARY OUTCOMES:
Impact of optimizing indocyanine green (ICG) dosage and storage conditions on total procedural cost. | Baseline (pre-procedure) and up to 24 weeks post-procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Bedynska M, Szewczyk G, Klepacka T, Sachadel K, Maciejewski T, Szukiewicz D, Fijalkowska A. Sentinel lymph node mapping using indocyanine green in patients with uterine and cervical neoplasms: restrictions of the method. Arch Gynecol Obstet. 2019 May;299(5):1373-1384. doi: 10.1007/s00404-019-05063-6. Epub 2019 Feb 14. PMID 30762108
- [Background] Laufer J, Scasso S, Papadia A. Impact of Indocyanine Green Dose on Sentinel Lymph Node Mapping in Cervical Cancer: A Systematic Review. Cancers (Basel). 2024 Sep 8;16(17):3107. doi: 10.3390/cancers16173107. PMID 39272965
- [Background] Cibula D, Potter R, Planchamp F, Avall-Lundqvist E, Fischerova D, Haie Meder C, Kohler C, Landoni F, Lax S, Lindegaard JC, Mahantshetty U, Mathevet P, McCluggage WG, McCormack M, Naik R, Nout R, Pignata S, Ponce J, Querleu D, Raspagliesi F, Rodolakis A, Tamussino K, Wimberger P, Raspollini MR. The European Society of Gynaecological Oncology/European Society for Radiotherapy and Oncology/European Society of Pathology Guidelines for the Management of Patients With Cervical Cancer. Int J Gynecol Cancer. 2018 May;28(4):641-655. doi: 10.1097/IGC.0000000000001216. PMID 29688967
- [Background] Abu-Rustum N, Yashar C, Arend R, Barber E, Bradley K, Brooks R, Campos SM, Chino J, Chon HS, Chu C, Crispens MA, Damast S, Fisher CM, Frederick P, Gaffney DK, Giuntoli R, Han E, Holmes J, Howitt BE, Lea J, Mariani A, Mutch D, Nagel C, Nekhlyudov L, Podoll M, Salani R, Schorge J, Siedel J, Sisodia R, Soliman P, Ueda S, Urban R, Wethington SL, Wyse E, Zanotti K, McMillian NR, Aggarwal S. Uterine Neoplasms, Version 1.2023, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2023 Feb;21(2):181-209. doi: 10.6004/jnccn.2023.0006. PMID 36791750